CLINICAL TRIAL: NCT03734783
Title: Regulate Effect of Il-35 Secreting Breg Cells on Tcells and on Diseases Progression in Patients With CHB
Brief Title: IL-35+Breg/Il-35 Effect on T Cell Immune in Patients With CHB
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, LiangXS, Professor, Changhai Hospital
Other Study IDs: 16ZR1400400
Record Dates: First submitted 2018-10-31; First posted 2018-11-08 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Chronic Hepatitis b
Keywords: chronic hepatitis B; regulating B cells; T help 17 cells; Interleukin 35
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: HBsAg positive more than 6 months
- health control

SUMMARY:
The investigators observed the level of IL-35 secreting B regulatory (IL-35+Bregs) cells in peripheral blood cells in patients with chronic hepatitis B, and analysed the relationship between the IL-35+Bregs level and disease stage, and Th1 and Th2 cells level.

DETAILED DESCRIPTION:
Regulatory B cells (Bregs) are involved in the immune tolerance process through multiple pathways and Bregs are involved in the process of chronic HBV infection.

Here the investigators intended to investigate the regulating role and the mechanism of CD19+ IL-35+ cells on host T cell immune during chronic HBV infection by using in vitro cell sorting, B cell differentiation induction, Transwell cell co-culture system and other methods.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic hepatitis B virus infection
* 17<age<70
* Can read, understand and sign patients informed consent

Exclusion Criteria:

* Co-infection with HCV,HIV,HDV etc.
* Have malignancy
* Have uncontrollable extra-hepatic disease

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic hepatitis B infection
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
IL-35+Bregs level | ENROLLED DAY
  IL-35 secreting regulatory B cells level in patients with CHB
IL-35+Bregs regulatory effect | enrolled day
  regulatory effect of IL-35+Bregs on T cell immune

SECONDARY OUTCOMES:
IL-35+Bregs phenotype | enrolled day
  the main phenotype of IL-35 secreting Bregs

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai hospital, Shanghai, China

REFERENCES:
- [Derived] Liu Y, Luo Y, Zhu T, Jiang M, Tian Z, Tang G, Liang X. Regulatory B Cells Dysregulated T Cell Function in an IL-35-Dependent Way in Patients With Chronic Hepatitis B. Front Immunol. 2021 Apr 12;12:653198. doi: 10.3389/fimmu.2021.653198. eCollection 2021. PMID 33912178